CLINICAL TRIAL: NCT04640883
Title: Effects of Including 30-s Sprints During Low-intensity Cycling Exercises During a Training Camp on Performance and Muscle/Blood Characterisitcs
Brief Title: Effects of Including Sprints During Low-intensity Cycling Exercises on Performance and Muscle/Blood Characteristics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Trainome 2017#011
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Healthy; Cyclists
Keywords: Sprint; Low-intensity cycling; Skeletal muscle; Endurance performance
MeSH Terms: interventions — Salvage Therapy

STUDY DESIGN:
Intervention Model Description: Investigating the effects of including sprints during low-intensity training sessions during a 14-d training camp with increased training load on performance and muscle/blood biology
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprints during low-intensity cycling (Experimental)
  Interventions: Behavioral: Inclusion of sprints during low-intensity cycling during a 14-day training camp (high training load); Behavioral: Recovery for 10 days (low training load)
- Low-intensity cycling (Active Comparator)
  Interventions: Behavioral: Low-intensity cycling during a 14-day training camp (high training load); Behavioral: Recovery for 10 days (low training load)

INTERVENTIONS:
Behavioral: Inclusion of sprints during low-intensity cycling during a 14-day training camp (high training load) — Inclusion of 12x30-s maximal sprints during five low-intensity cycling sessions with long duration (>fours hours per session). Five sessions will be performed as low-intensity cycling-only (Controll sessions, distance matched). All other sessions will be performed as low-intensity sessions and adjusted according to each participants training load goal to reach an increase of ~50% in load compared to habitual training.
  Arms: Sprints during low-intensity cycling
Behavioral: Low-intensity cycling during a 14-day training camp (high training load) — Five low-intensity cycling sessions (>four hours per session), distance-matched to sprint group.
  Arms: Low-intensity cycling
Behavioral: Recovery for 10 days (low training load) — Habitual low-intensity cycling (>0.5-2 hours per session)

SUMMARY:
To investigate the effects of Including 30-s sprints during low-intensity cycling exercises during a training camp on performance and muscle/blood characterisitcs in elite cyclists

DETAILED DESCRIPTION:
Inclusion of sprint intervals during low-intensity training (LIT) sessions has been suggested as a potential mean to improve endurance performance in elite cyclists, facilitated by muscular or systemic physiological adaptations. So far, the effects of such training has been studied exclusively in context of short-lasting low-intensity sessions, representing a scenario with suboptimal ecological validity for such highly trained athetes.

This study will investigate the effects of including sprints during prolonged LIT-sessions sessions during a 14-day training camp focusing on LIT, followed by 10 days recovery (REC), on performance and performance-related measures in elite cyclists. During the training camp, a sprint training group will conduct 12x30-s maximal sprints during five LIT sessions, whereas a control group will perform distance-matched LIT-only. Overall, the training camp will lead to substantial increases in training load compared to habitual training in both intervention groups, followed by subsequent reductions during REC. Performance tests will be conducted before the training camp (T0) and after REC (T2). Muscle biopsies, hematological measures and stress/recovery questionnaires will be collected Pre (T0) and after the camp (T1).

The study was pre-registered at Norwegian Center for Research Data (14/08/2017, Norwegian): http://pvo.nsd.no/prosjekt/55322

ELIGIBILITY:
Inclusion Criteria:

* VO2max > 65ml/kg/min

Exclusion Criteria:

* VO2max < 65ml/kg/min
* Average endurance training per week >10hrs/wk during the four weeks leading up to the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2017-12-23 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
Performance during a 5-minute all-out cycling test | Changes from before the intervention (T0) to immediately after the intervention (T2, after REC)
  Mean power output measured during a 5-minute all-out cycling test performed at the end of a ~2 hour long exercise protocol

SECONDARY OUTCOMES:
Sprint performance | Changes from before the intervention (T0) to immediately after the intervention (T2, after REC)
  Mean power output measured during four consecutive 30-s maximal sprints
Maximal oxygen uptake | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Maximal oxygen consumption measured during an incremental cycling exercise test to exhaustion
Maximal aerobic power output | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Maximal aerobic power output measured as mean power output during the last minute of an incremental cycling exercise test to exhaustion
Gross efficiency (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Contribution of total energy turnover to power output in the fresh and fatigued state incremental cycling exercise test (with 5 minute steps)
Gross efficiency (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Contribution of total energy turnover to power output in the fresh and fatigued state incremental cycling exercise test (with 5 minute steps)
Power output at lactate threshold (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Power output at 4 mmol blood lactate concentration measured during an incremental cycling exercise test (with 5 minute steps)
Power output at lactate threshold (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Power output at 4 mmol blood lactate concentration measured during an incremental cycling exercise test (with 5 minute steps)
Fractional utilization of VO2max (incremental test) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Fractional utilization of VO2max measured at 4 mmol blood lactate concentrations measured during an incremental cycling exercise test (with 5 minute steps)
Fractional utilization of VO2max (5-min test) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Fractional utilization of VO2max measured during the 5-min test
Protein abundance in skeletal muscle | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Protein abundances in m. vastus lateralis measured using western blotting
Haemoglobin mass (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Hemoglobin mass measured using CO rebreathing (g)
Haemoglobin mass (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Hemoglobin mass measured using CO rebreathing (g)
Blood volume (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Blood volume measured using CO rebreathing
Blood volume (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Blood volume measured using CO rebreathing
Plasma volume (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Plasma volume measured using CO rebreathing
Plasma volume (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Plasma volume measured using CO rebreathing
Red blood cell volume (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Red blood cell volume measured using CO rebreathing
Red blood cell volume (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Red blood cell volume measured using CO rebreathing
Mean corposcular volume (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Mean corposcular volume measured using CO rebreathing
Mean corposcular volume (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Mean corposcular volume measured using CO rebreathing
Hematocrit (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Hematocrit measured using centrifugation
Hematocrit (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Hematocrit measured using centrifugation
Body mass (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Body mass (kg) measured using Dual-energy X-ray absorptiometry
Body mass (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Body mass (kg) measured using Dual-energy X-ray absorptiometry
Enzyme activity in skeletal muscle | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Enzyme activity in m. vastus lateralis measured using ELISA kits (I.e., CS and PFK)
Lean body mass (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Lean body mass (kg) measured using Dual-energy X-ray absorptiometry
Lean body mass (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Lean body mass (kg) measured using Dual-energy X-ray absorptiometry
Fat mass (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Fat mass (kg) measured using Dual-energy X-ray absorptiometry
Fat mass (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Fat mass (kg) measured using Dual-energy X-ray absorptiometry
Session rate of percieved exertion | Throughout the training camp (14 days)
  Session rate of percieved exertion (sRPE) measured after each exercise involving sprints/control exercise using a 9-point scale ranging from "very, very demotivated" to "very, very motivated" (1 to 9)
Stress-recovery state (training camp) | Changes from before the intervention (T0) to immediately after the training camp (T1)
  Recovery state of participants measured using Recovery-Stress Questionnaire for Athletes (RESTQ-36-R-Sport, 36 questions, 7-point scale ranging from 0/never to 6/always)
Stress-recovery state (recovery/REC) | Changes from before the intervention (T0) to immediately after the intervention (T2, i.e. after REC)
  Recovery state of participants measured using Recovery-Stress Questionnaire for Athletes (RESTQ-36-R-Sport, 36 questions, 7-point scale ranging from 0/never to 6/always)

OTHER OUTCOMES:
Training load | From four weeks prior to the intervention and throughout the study, an average of 52 days
  Training load calculated as time spent in different heart rate zones using the individualized TRIMP method

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Lofthus, Study Chair — Research Administrator
Locations (1):
- Inland Norway University of Applied Sciences, Lillehammer, Norway

REFERENCES:
- [Background] Almquist NW, Ellefsen S, Sandbakk O, Ronnestad BR. Effects of including sprints during prolonged cycling on hormonal and muscular responses and recovery in elite cyclists. Scand J Med Sci Sports. 2021 Mar;31(3):529-541. doi: 10.1111/sms.13865. Epub 2020 Nov 7. PMID 33113253
- [Background] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482
- [Background] Sylta O, Tonnessen E, Seiler S. From heart-rate data to training quantification: a comparison of 3 methods of training-intensity analysis. Int J Sports Physiol Perform. 2014 Jan;9(1):100-7. doi: 10.1123/IJSPP.2013-0298. PMID 24408353
- [Background] Manzi V, Iellamo F, Impellizzeri F, D'Ottavio S, Castagna C. Relation between individualized training impulses and performance in distance runners. Med Sci Sports Exerc. 2009 Nov;41(11):2090-6. doi: 10.1249/MSS.0b013e3181a6a959. PMID 19812506
- [Background] Almquist NW, Ettema G, Hopker J, Sandbakk O, Ronnestad BR. The Effect of 30-Second Sprints During Prolonged Exercise on Gross Efficiency, Electromyography, and Pedaling Technique in Elite Cyclists. Int J Sports Physiol Perform. 2019 Nov 5;15(4):562-570. doi: 10.1123/ijspp.2019-0367. Print 2020 Apr 1. PMID 31693997
- [Background] Siebenmann C, Robach P, Jacobs RA, Rasmussen P, Nordsborg N, Diaz V, Christ A, Olsen NV, Maggiorini M, Lundby C. "Live high-train low" using normobaric hypoxia: a double-blinded, placebo-controlled study. J Appl Physiol (1985). 2012 Jan;112(1):106-17. doi: 10.1152/japplphysiol.00388.2011. Epub 2011 Oct 27. PMID 22033534
- [Background] Thomsen JK, Fogh-Andersen N, Bulow K, Devantier A. Blood and plasma volumes determined by carbon monoxide gas, 99mTc-labelled erythrocytes, 125I-albumin and the T 1824 technique. Scand J Clin Lab Invest. 1991 Apr;51(2):185-90. doi: 10.1080/00365519109091106. PMID 2042022
- [Background] Almquist NW, Lovlien I, Byrkjedal PT, Spencer M, Kristoffersen M, Skovereng K, Sandbakk O, Ronnestad BR. Effects of Including Sprints in One Weekly Low-Intensity Training Session During the Transition Period of Elite Cyclists. Front Physiol. 2020 Sep 11;11:1000. doi: 10.3389/fphys.2020.01000. eCollection 2020. PMID 33041839
- [Background] Foster C. Monitoring training in athletes with reference to overtraining syndrome. Med Sci Sports Exerc. 1998 Jul;30(7):1164-8. doi: 10.1097/00005768-199807000-00023. PMID 9662690
- [Background] Borg G, Hassmen P, Lagerstrom M. Perceived exertion related to heart rate and blood lactate during arm and leg exercise. Eur J Appl Physiol Occup Physiol. 1987;56(6):679-85. doi: 10.1007/BF00424810. PMID 3678222
- [Background] Meinild Lundby AK, Jacobs RA, Gehrig S, de Leur J, Hauser M, Bonne TC, Fluck D, Dandanell S, Kirk N, Kaech A, Ziegler U, Larsen S, Lundby C. Exercise training increases skeletal muscle mitochondrial volume density by enlargement of existing mitochondria and not de novo biogenesis. Acta Physiol (Oxf). 2018 Jan;222(1). doi: 10.1111/apha.12905. Epub 2017 Jul 6. PMID 28580772
- [Background] Hopkins WG, Marshall SW, Batterham AM, Hanin J. Progressive statistics for studies in sports medicine and exercise science. Med Sci Sports Exerc. 2009 Jan;41(1):3-13. doi: 10.1249/MSS.0b013e31818cb278. PMID 19092709
- [Background] Fernandez-Garcia B, Perez-Landaluce J, Rodriguez-Alonso M, Terrados N. Intensity of exercise during road race pro-cycling competition. Med Sci Sports Exerc. 2000 May;32(5):1002-6. doi: 10.1097/00005768-200005000-00019. PMID 10795793
- [Background] Menaspa P, Quod M, Martin DT, Peiffer JJ, Abbiss CR. Physical Demands of Sprinting in Professional Road Cycling. Int J Sports Med. 2015 Nov;36(13):1058-62. doi: 10.1055/s-0035-1554697. Epub 2015 Aug 7. PMID 26252551
- [Background] Joyner MJ, Coyle EF. Endurance exercise performance: the physiology of champions. J Physiol. 2008 Jan 1;586(1):35-44. doi: 10.1113/jphysiol.2007.143834. Epub 2007 Sep 27. PMID 17901124
- [Background] Jeukendrup AE, Craig NP, Hawley JA. The bioenergetics of World Class Cycling. J Sci Med Sport. 2000 Dec;3(4):414-33. doi: 10.1016/s1440-2440(00)80008-0. PMID 11235007
- [Background] Padilla S, Mujika I, Cuesta G, Goiriena JJ. Level ground and uphill cycling ability in professional road cycling. Med Sci Sports Exerc. 1999 Jun;31(6):878-85. doi: 10.1097/00005768-199906000-00017. PMID 10378916
- [Background] Faria EW, Parker DL, Faria IE. The science of cycling: physiology and training - part 1. Sports Med. 2005;35(4):285-312. doi: 10.2165/00007256-200535040-00002. PMID 15831059
- [Background] Zapico AG, Calderon FJ, Benito PJ, Gonzalez CB, Parisi A, Pigozzi F, Di Salvo V. Evolution of physiological and haematological parameters with training load in elite male road cyclists: a longitudinal study. J Sports Med Phys Fitness. 2007 Jun;47(2):191-6. PMID 17557057
- [Background] Lucia A, Chicharro JL, Perez M, Serratosa L, Bandres F, Legido JC. Reproductive function in male endurance athletes: sperm analysis and hormonal profile. J Appl Physiol (1985). 1996 Dec;81(6):2627-36. doi: 10.1152/jappl.1996.81.6.2627. PMID 9018515
- [Background] Lucia A, Hoyos J, Pardo J, Chicharro JL. Metabolic and neuromuscular adaptations to endurance training in professional cyclists: a longitudinal study. Jpn J Physiol. 2000 Jun;50(3):381-8. doi: 10.2170/jjphysiol.50.381. PMID 11016988
- [Background] Hawley JA, Stepto NK. Adaptations to training in endurance cyclists: implications for performance. Sports Med. 2001;31(7):511-20. doi: 10.2165/00007256-200131070-00006. PMID 11428688
- [Background] Saw AE, Halson SL, Mujika I. Monitoring Athletes during Training Camps: Observations and Translatable Strategies from Elite Road Cyclists and Swimmers. Sports (Basel). 2018 Jul 20;6(3):63. doi: 10.3390/sports6030063. PMID 30036955
- [Background] Costill DL, Thomas R, Robergs RA, Pascoe D, Lambert C, Barr S, Fink WJ. Adaptations to swimming training: influence of training volume. Med Sci Sports Exerc. 1991 Mar;23(3):371-7. PMID 2020277
- [Background] Bellinger P. Functional Overreaching in Endurance Athletes: A Necessity or Cause for Concern? Sports Med. 2020 Jun;50(6):1059-1073. doi: 10.1007/s40279-020-01269-w. PMID 32064575
- [Background] Slivka DR, Hailes WS, Cuddy JS, Ruby BC. Effects of 21 days of intensified training on markers of overtraining. J Strength Cond Res. 2010 Oct;24(10):2604-12. doi: 10.1519/JSC.0b013e3181e8a4eb. PMID 20733522
- [Background] Halson SL, Bridge MW, Meeusen R, Busschaert B, Gleeson M, Jones DA, Jeukendrup AE. Time course of performance changes and fatigue markers during intensified training in trained cyclists. J Appl Physiol (1985). 2002 Sep;93(3):947-56. doi: 10.1152/japplphysiol.01164.2001. PMID 12183490
- [Background] Jeukendrup AE, Hesselink MK, Snyder AC, Kuipers H, Keizer HA. Physiological changes in male competitive cyclists after two weeks of intensified training. Int J Sports Med. 1992 Oct;13(7):534-41. doi: 10.1055/s-2007-1021312. PMID 1459749
- [Background] Le Meur Y, Pichon A, Schaal K, Schmitt L, Louis J, Gueneron J, Vidal PP, Hausswirth C. Evidence of parasympathetic hyperactivity in functionally overreached athletes. Med Sci Sports Exerc. 2013 Nov;45(11):2061-71. doi: 10.1249/MSS.0b013e3182980125. PMID 24136138
- [Background] Le Meur Y, Louis J, Aubry A, Gueneron J, Pichon A, Schaal K, Corcuff JB, Hatem SN, Isnard R, Hausswirth C. Maximal exercise limitation in functionally overreached triathletes: role of cardiac adrenergic stimulation. J Appl Physiol (1985). 2014 Aug 1;117(3):214-22. doi: 10.1152/japplphysiol.00191.2014. Epub 2014 Jun 12. PMID 24925979
- [Background] Valstad SA, von Heimburg E, Welde B, van den Tillaar R. Comparison of Long and Short High-Intensity Interval Exercise Bouts on Running Performance, Physiological and Perceptual Responses. Sports Med Int Open. 2017 Dec 18;2(1):E20-E27. doi: 10.1055/s-0043-124429. eCollection 2018 Jan. PMID 30539113
- [Background] Laursen PB, Shing CM, Peake JM, Coombes JS, Jenkins DG. Interval training program optimization in highly trained endurance cyclists. Med Sci Sports Exerc. 2002 Nov;34(11):1801-7. doi: 10.1097/00005768-200211000-00017. PMID 12439086
- [Background] MacDougall JD, Hicks AL, MacDonald JR, McKelvie RS, Green HJ, Smith KM. Muscle performance and enzymatic adaptations to sprint interval training. J Appl Physiol (1985). 1998 Jun;84(6):2138-42. doi: 10.1152/jappl.1998.84.6.2138. PMID 9609810
- [Background] Gunnarsson TP, Brandt N, Fiorenza M, Hostrup M, Pilegaard H, Bangsbo J. Inclusion of sprints in moderate intensity continuous training leads to muscle oxidative adaptations in trained individuals. Physiol Rep. 2019 Feb;7(4):e13976. doi: 10.14814/phy2.13976. PMID 30793541
- [Background] Hostrup M, Bangsbo J. Limitations in intense exercise performance of athletes - effect of speed endurance training on ion handling and fatigue development. J Physiol. 2017 May 1;595(9):2897-2913. doi: 10.1113/JP273218. Epub 2016 Nov 16. PMID 27673449
- [Background] Skovgaard C, Almquist NW, Kvorning T, Christensen PM, Bangsbo J. Effect of tapering after a period of high-volume sprint interval training on running performance and muscular adaptations in moderately trained runners. J Appl Physiol (1985). 2018 Feb 1;124(2):259-267. doi: 10.1152/japplphysiol.00472.2017. Epub 2017 Sep 21. PMID 28935825
- [Background] Skovgaard C, Brandt N, Pilegaard H, Bangsbo J. Combined speed endurance and endurance exercise amplify the exercise-induced PGC-1alpha and PDK4 mRNA response in trained human muscle. Physiol Rep. 2016 Jul;4(14):e12864. doi: 10.14814/phy2.12864. PMID 27456910
- [Background] Brandt N, Gunnarsson TP, Hostrup M, Tybirk J, Nybo L, Pilegaard H, Bangsbo J. Impact of adrenaline and metabolic stress on exercise-induced intracellular signaling and PGC-1alpha mRNA response in human skeletal muscle. Physiol Rep. 2016 Jul;4(14):e12844. doi: 10.14814/phy2.12844. PMID 27436584
- [Background] Sjogaard G. Muscle morphology and metabolic potential in elite road cyclists during a season. Int J Sports Med. 1984 Oct;5(5):250-4. doi: 10.1055/s-2008-1025915. PMID 6500791
- [Background] Coyle EF, Feltner ME, Kautz SA, Hamilton MT, Montain SJ, Baylor AM, Abraham LD, Petrek GW. Physiological and biomechanical factors associated with elite endurance cycling performance. Med Sci Sports Exerc. 1991 Jan;23(1):93-107. PMID 1997818